CLINICAL TRIAL: NCT06441695
Title: The Acute Effects of PLT Health Solutions zümXR Extended-Release Caffeine on Side Effects, Mood and Alertness Following a Night of Suboptimal Sleep
Brief Title: Acute Effects of PLT Health Solutions zümXR Extended-Release Caffeine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00078903
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Caffeine; Cognitive Change; Mood; Mood Change
Keywords: extended release caffeine; caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Treatment (Experimental): extended release xumXR caffeine (200mg) capsule; subject receives 2 capsules totaling 400mg
  Interventions: Dietary Supplement: xumXR extended release caffeine
- Control Treatment (Active Comparator): immediate release caffeine (200mg) capsule; subject receives 2 capsules totaling 400mg
  Interventions: Dietary Supplement: immediate release caffeine

INTERVENTIONS:
Dietary Supplement: xumXR extended release caffeine — proprietary capsule for extended release of caffeine
  Arms: Experimental Treatment
Dietary Supplement: immediate release caffeine — immediate release caffeine capsule
  Arms: Control Treatment

SUMMARY:
This will be a (2 visit) double-blind, randomized, crossover design clinical study to assess the potential benefits of ER-CAFF versus IR-CAFF by assessing its impact on side effect profiles, mood states, alertness, and cognitive abilities following ingestion after a suboptimal night of sleep. This study will enroll 30 healthy men and women who will be recruited by word of mouth, email contact, and direct contact from the greater Tampa Bay Area. To account for potential dropouts, we aim to enroll approximately 20% over the desired sample size (total of 36 participants). The anticipated study period will last approximately 2 weeks.

After initial pre-screening, participants will report to the laboratory on two separate occasions after an overnight fast (10 hours minimum). Participants will be required to have a night of partial sleep deprivation the night before (<5 hours sleep), which will be confirmed by self reported sleep logs and objective multisensor (triaxial accelerometry and cardiac data) wearable devices to accurately measure sleep deficit data. Upon arrival, participants will undergo baseline (BL) testing and then ingest a bolus of one study product with 4-8 ounces of water: 400 mg zümXR extended-release caffeine (ER-CAFF), or 400 mg of immediate-release caffeine anhydrous (IR-CAFF) (2 group, crossover design). Thereafter, participants will undergo subsequent testing sessions at 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation. After the 4-hour (240 min) measurements, a caffeine-free food bar will be provided. This same food bar will also be offered to participants following the final 7-hour (420 min) measurements. The precise measures and timepoints for the measures are further defined below. There will be a one-week minimum washout period between treatments in the crossover design.

DETAILED DESCRIPTION:
Pre-screening/enrollment (Day -30 to Day -1) The potential subject will present a health history / Caffeine Consumption / Morningness-Eveningness questionnaires to screen for study eligibility described in sections 5.2.1 (inclusion criteria) and 5.2.2 (exclusion criteria). The questionnaires will be reviewed by the Investigator or designee. If the subject is eligible, they will be contacted by phone to walk through the study requirements and answer any questions. If the subject qualifies and is amenable with the study requirements, we will obtain written consent via an IRB approved ICF. The potential subject will be given the opportunity to review the ICF, ask any questions they may have to the Investigator or designee. The potential subject will be required to sign the ICF for study enrollment and to proceed with study participation.

Baseline assessment (Day 0, Visit 1) After initial pre-screening, participants will report to the laboratory on two separate occasions after an overnight fast (10 hours minimum). Participants will be required to have a night of partial sleep deprivation the night before (≤ 5 hours sleep), which will be confirmed by self reported sleep logs and objective multisensor (triaxial accelerometry and cardiac data) wearable devices to accurately measure sleep deficit data (Roberts et al., 2020). Upon arrival, participants will undergo baseline (BL) testing (Heart rate, blood pressure, Caffeine VAS, Samn-Perilli/Thayer's, PANAS, PVT, RVIP). Immediately after, subjects will ingest a bolus of one study product (either ER-CAFF or IR-CAFF) with 4-8 ounces of water: 400 mg zümXR extended-release caffeine (ER-CAFF), or 400 mg of immediate-release caffeine (IR-CAFF) (2 group, crossover design). Thereafter, participants will undergo subsequent testing sessions at 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation. This testing will include the vitals listed above, a subset of the BL tests according to the time point (see below, Table 2), and queried about adverse events. At the 4-hour (240 min) measurement, a standardized caffeine-free food bar will be provided. This food bar will also be offered to participants following the final 7-hour (420 min) measurements. After the completion of Day 0, There will be a one-week minimum washout period between treatments in the crossover design.

Final Testing (Day 1, Visit 2):

After the one-week minimum washout period, subjects will report back to the lab and will repeat Day 0 testing with the other supplement (either ER-CAFF or IR-CAFF). Following this testing, the subjects will have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 35-50 years (both limits inclusive);
* Body mass index (BMI) of 18.50-29.99 kg/m2 -Habitual moderate caffeine consumers (200-400 mg/day) assessed through caffeine assessment tool (Caffeine -
* Consumption Questionnaire, CCQ);
* Intermediate chronotype (>31 or <69 on Morningness-Eveningness Questionnaire).

Exclusion Criteria:

* Subjects presenting any of the following will not be included in the study:
* No history of anxiety disorders or sleep disorders;
* Non-smokers;
* Alcohol consumption 72 hours prior to the start of study/consumption of study product;
* No use of sleep medicines, melatonin, marijuana within two weeks of start of study;
* No travel involving time zone change, shift work, or other life events that alter sleep schedule >3 hours from the norm one week before the start of study (assessed using sleep-wake schedule diary for week prior to study);
* Caffeine restricted past 12 PM from the day prior to the start of study (verify through caffeine diet history).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Changes in Concentration using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Higher values indicate greater alertness and is considered to be a better outcome.
Changes in Energy using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Higher values indicate greater energy and is considered to be a better outcome.
Changes in Confidence using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Higher values indicate greater energy and is considered to be a better outcome.
Changes in Mood Enhancement using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Higher values indicate greater mood enhancements and is considered to be a better outcome.
Changes in Jitteriness using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Lower values indicate less jitters and is considered to be a better outcome.
Changes in Anxiousness using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Lower values indicate less jitters and is considered to be a better outcome.
Changes in Sleepy using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Lower values indicate less jitters and is considered to be a better outcome.
Changes in Irritability using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Lower values indicate less jitters and is considered to be a better outcome.
Changes in Heart Rate (Heart Pounding) using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Lower values indicate less jitters and is considered to be a better outcome.
Changes in Headache using Visual Analog Scale (VAS) | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  The test consists of a horizontal line, with endpoints labeled as "no effect" or "extremely high effect" to represent the continuum of caffeine effects experienced by the subject. Users mark on the line to indicate their perception regarding caffeine effects. Scoring is from 0 (no effect) to 100 (extremely high effect). Lower values indicate less jitters and is considered to be a better outcome.
Heart rate (HR) | baseline, 45, 60, 135, 240, 360, and 420 minutes post-supplementation
  Changes in heart rate post supplementation; resting HR measured using pulse oximeter
Diastolic blood pressure (BP) | baseline, 45, 60, 135, 240, 360, and 420 minutes post-supplementation
  Changes in diastolic BP post supplementation. Resting blood pressure measured using an automated BP cuff.
Systolic blood pressure (BP) | baseline, 45, 60, 135, 240, 360, and 420 minutes post-supplementation
  Changes in systolic BP post supplementation. Resting blood pressure measured using an automated BP cuff.

SECONDARY OUTCOMES:
Changes in Rapid Visual Information Processing | baseline , 90 and 300 minutes post-supplementation.
  This 12 minute test checks how well you can quickly spot specific patterns on a screen, helping measure your attention and focus. A participant is presented with a series of digits (1-9) on a computer screen. The presentation time is 100 digits/min (or 1digit/600ms). The participant's task is to press a response key (here: Spacebar) as soon as she detects a series of three consecutive odd or three consecutive even digits.
Changes in Psychomotor Vigilance Test | baseline , 90 and 300 minutes post-supplementation.
  This test measures how quickly and accurately you can respond to simple tasks, like pressing a button when you see a specific symbol. It assesses your reaction time and attention span. Participants are instructed to press the <Spacebar> as fast as possible after a red stopwatch appears on screen. A valid response (response occurs after a stopwatch appears) is followed by reaction time feedback.
Changes in Samn-Perelli/Thayer's scale (aka Stanford Sleepiness Scale) | baseline, 90, 300, and 420 minutes post-supplementation.
  This subjective assessment tool will be used to measure the subject's perceived level of sleepiness or alertness. This tool consists of seven statements or descriptions, each corresponding to a different level of sleepiness or alertness. Respondents are asked to select the statement that best describes their current level of alertness. The scale ranges from 1 to 7, with 1 indicating the highest level of alertness (feeling active, vital, alert, or wide awake) and 7 indicating the lowest level of alertness (no longer fighting sleep, sleep onset soon, having dream-like thoughts).
Changes in Positive & Negative Affect Schedule (PANAS) | baseline, 90, 300, and 420 minutes post-supplementation.
  This scale consists of a number of words that describe different feelings and emotions. Subject will choose a number 1 through 5 (1=Very slightly or not at all, 5=extremely) to describe the feeling/emotion listed. Overall positive and negative scores will be tallied for interpretation.

OTHER OUTCOMES:
Adverse Events | baseline, 45, 60, 90, 135, 240, 300, 360, and 420 minutes post-supplementation.
  Will be recorded based on observation and verbal subject questioning.
  Defined as participants self-reported adverse effects. Items that will be surveyed are headache, dizziness, nausea, vomiting, indigestion, blurred vision, lethargy, swelling, itching, chest pain, heart palpitations, difficulty breathing, lethargy, and muscle cramps.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Science & Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No